CLINICAL TRIAL: NCT02670967
Title: Effects of Soluble Fiber on Blood Pressure: A Meta-analysis of Randomly-controlled Trials
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: FIberBPMeta
Record Dates: First submitted 2015-08-11; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Soluble Fibre

SUMMARY:
The present study conducted a meta-analysis of 22 randomly controlled trials to assess the effects of soluble fiber intake on blood pressure in human subjects.

Using the Cochrane Handbook for Systematic Reviews of Intervention, a systematic review and meta-analysis was conducted. Information regarding study methods, characteristics, mean BP and standard deviations were extracted The data from each study were pooled using a random effects model to estimate the effects of soluble fiber consumption on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Randomized Controlled Trials
* Parallel or Crossover Design
* Duration: >3 weeks
* Human trials
* Viscous (soluble) fiber
* Viable endpoint data
* Articles published in English

Exclusion Criteria:

* Non-human
* Non-randomized
* Lack of control
* Less than 4 weeks in duration
* No viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy, hypertensive, hypercholesterolaemic, diabetic
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 4 weeks
Diastolic Blood Pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto; Kashif Khan, BSc, Study Director — Unity Health Toronto
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Khan K, Jovanovski E, Ho HVT, Marques ACR, Zurbau A, Mejia SB, Sievenpiper JL, Vuksan V. The effect of viscous soluble fiber on blood pressure: A systematic review and meta-analysis of randomized controlled trials. Nutr Metab Cardiovasc Dis. 2018 Jan;28(1):3-13. doi: 10.1016/j.numecd.2017.09.007. Epub 2017 Oct 7. PMID 29153856